CLINICAL TRIAL: NCT06775717
Title: Comparative Effects of Motor Imagery and Mirror Therapy on Synkinesis, Facial Asymmetry, Facial Function and Quality of Life in Bell's Palsy Patients.
Brief Title: Motor Imagery and Mirror Therapy on Synkinesis, Facial Asymmetry, Facial Function and QoF in Bell's Palsy Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: REC\RCR & AHS\24\0252
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Bell Palsy
Keywords: Facial asymmetry; Quality of life; Facial function; Mirror therapy; Motor Imagery
MeSH Terms: conditions — Bell Palsy; Facial Asymmetry | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery with conventional Treatment. (Experimental): 21 patients will get the mirror therapy. Duration of sessions will be 35 minutes, with 5 sessions a week in 4 weeks.
  Interventions: Other: Motor Imagery with conventional Treatment; Other: Mirror therapy with conventional Treatment.
- Mirror therapy with conventional Treatment. (Active Comparator): 21 patients will get the mirror therapy. Duration of sessions will be 35 minutes, with 5 sessions a week in 4 consecutive weeks.
  Interventions: Other: Motor Imagery with conventional Treatment; Other: Mirror therapy with conventional Treatment.

INTERVENTIONS:
Other: Motor Imagery with conventional Treatment — This treatment will be given 5 sessions a week in 4 consecutive weeks.
Other: Mirror therapy with conventional Treatment. — This treatment will be given 5 sessions a week in 4 consecutive weeks.

SUMMARY:
Bell's palsy is a condition that causes sudden weakness in the muscles on one side of the face. The weakness makes half of the face appear to droop, difficulty in closing eyes and synkinesis. Mirror therapy and Motor imagery have shown promise in improving motor function and overall well-being.

Participant will be assigned two groups, A and B. All the groups will receive interventions for five days a week for 8 weeks and treatment time will be 35 minutes. The outcome measuring scales used will be facial Clinometric Scale (FaCE), Synkinesis Assessment Scale and Sunnybrook facial grading system to assess facial symmetry, synkinesis and facial movements, data will be collected on SPSS.

DETAILED DESCRIPTION:
Bell's palsy is a condition that causes sudden weakness in the muscles on one side of the face. The weakness makes half of the face appear to droop, difficulty in closing eyes and synkinesis. These symptoms significantly impact facial symmetry and quality of life. Mirror therapy and Motor imagery have shown promise in improving motor function and overall well-being. The primary objective of this study is to compare the effects of the Mirror therapy and Motor Imagery on facial symmetry, synkinesis and quality of life in patients with Bell's palsy. This randomized clinical trial will be carried in 10 months after the approval of synopsis. Total number of 36 participants meeting the inclusion criteria will be included in this study through a non-probability convenience sampling technique. Participants will be randomly assigned into 2 groups using computer generated randomization method. Group A and Group participants will receive Motor Imagery and Mirror therapy, respectively. All the groups will receive interventions for five days a week for 8 weeks. Total treatment time will be 35 minutes. The outcome measuring scales used will be facial Clinometric Scale (FaCE), Synkinesis Assessment Scale and Sunnybrook facial grading system to assess facial symmetry, synkinesis and facial movements. The data will be analyze using SPSS version 28 for windows. Assessment will be carried out at baseline and four weeks, after discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above.
* Both genders male and female will be included.
* Patients diagnosed with Bell's palsy with relevant diagnostic criteria, including history. (tick bite, erythema migraine, pain), neurological examination including inspection of ear and infection of HIV, Herpes virus.
* Patient having asymmetry in face (Sunnybrook Facial Grading Scale SFGS, use to check asymmetry in both sides of face).
* Appearance of synkinesis on affected side (Synkinesis Assessment Scale)
* Onset of symptoms must be first week.
* Patient having sufficient, physical, and mental ability to understand instructions and cooperate throughout the session.

Exclusion Criteria:

* Patients diagnosed with other than Bell's palsy (e.g., facial nerve trauma) (25).
* Patients with severe co-morbidities (e.g., uncontrolled hypertension, diabetes, cardiovascular diseases).
* Patients with significant cognitive impairment or communication difficulties who have undergone previous facial nerve surgery or interventions.
* Patients with severe psychiatric conditions affecting compliance or participation and on psychiatric medications.
* Patients with central nervous system tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The Facial Clinometric Scale: | 4 weeks
  The FaCE scale is a fascial palsy-related self-assessment QoL questionnaire comprising 15 questions based on a 5-point Likert-scale that evaluates the intensity and frequency of physical and psychosocial impairments in 6 domains of facial function: facial movement, facial comfort, eye comfort, oral function, lacrimal control and social function.
Sunnybrook Facial Grading Scale: | 4 weeks
  Sunnybrook scale is considered the current standard in evaluating outcomes and synkinesis due to its comprehensive scope, ease of use, and rapid results interpretation (27). The Sunnybrook facial grading scale, unlike others, systematically focuses on each subunit of facial movement (eyebrows, eyelids, nasal base, upper lip, and lower lip), while subjects are instructed to make six simple facial expressions.
Synkinesis Assessment Scale: | 4 weeks
  The phenomenon known as synkinesis occurs when there is intentional movement in one or more ipsilateral facial regions but involuntary movement in another area of the face.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Bashir Hospital., Sialkot, Punjab Province
  - Sulehri Children Hospital, Sialkot, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castaldo M, Sellitto G, Ruotolo I, Berardi A, Galeoto G. The Use of Mirror Therapy in Peripheral Seventh Nerve Palsy: A Systematic Review. Brain Sci. 2024 May 23;14(6):530. doi: 10.3390/brainsci14060530. PMID 38928530
- [Background] Patel H, Landge P, Barot J. A Comparative Study to Analyse the Effect of Motor Imagery and Mirror Book Therapy Versus Mime Therapy for the Recovery in Patients with Acute Bell's Palsy. Int J Sci Res. 2023;12(12):2047-55.
- [Background] Roh TS, Jung BK, Yun I, Lew DH, Kim YS. Effect of botulinum toxin A on vasoconstriction and sympathetic neurotransmitters in a murine random pattern skin flap model. Wound Repair Regen. 2017 Jan;25(1):75-85. doi: 10.1111/wrr.12501. Epub 2017 Jan 5. PMID 27997734
- [Background] Khanzada K, Ijaz Gondal M, Qamar M, Basharat A, Ahmad W, Ali S. Comparison of efficacy of Kabat rehabilitation and facial exercises along with nerve stimulation in patients with Bell's palsy. BLDE Univ J Heal Sci. 2018;3(1):31.
- [Background] Baugh RF, Basura GJ, Ishii LE, Schwartz SR, Drumheller CM, Burkholder R, Deckard NA, Dawson C, Driscoll C, Gillespie MB, Gurgel RK, Halperin J, Khalid AN, Kumar KA, Micco A, Munsell D, Rosenbaum S, Vaughan W. Clinical practice guideline: Bell's palsy. Otolaryngol Head Neck Surg. 2013 Nov;149(3 Suppl):S1-27. doi: 10.1177/0194599813505967. PMID 24189771
- [Background] Singh A, Deshmukh P. Bell's Palsy: A Review. Cureus. 2022 Oct 11;14(10):e30186. doi: 10.7759/cureus.30186. eCollection 2022 Oct. PMID 36397921